CLINICAL TRIAL: NCT07078279
Title: Evaluation of a Rehabilitation Intervention Using Immersive Virtual Reality to Improve Functional Balance in Children and Adolescents With Cerebral Palsy (GMFCS III-IV)
Brief Title: Effects of Virtual Reality on Functional Balance in Children With Cerebral Palsy (GMFCS III-IV)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartolome Puerta Arroyo (Other)
Collaborators: Rocío Martín Valero (Unknown)
Responsible Party: Sponsor-Investigator, Bartolome Puerta Arroyo, Doctorando Universidad Málaga, University of Malaga
Organization: University of Malaga (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04072025
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy; Functional Balance
Keywords: Functional balance; Cerebral palsy; Immersive virtual reality; Pediatric; Early Clinical Assessment of Balance (ECAB)
MeSH Terms: conditions — Cerebral Palsy | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Multicenter randomized clinical trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG): Intervention with Immersive Virtual Reality (VR) (Experimental): * Participants in the Experimental Group will receive a rehabilitation intervention focused on improving functional balance using immersive virtual reality (VR).
  * The intervention will be delivered using Meta Quest 3 headsets, a stand-alone, wireless, high-definition device that allows for a fully immersive experience.
  * Sessions will last 30 minutes, three times a week, for six weeks (total: 18 sessions).
  * Activities within the virtual environment are designed to promote:
  Postural control Static and dynamic balance Motor coordination
  * The physical therapist will supervise each session and adapt the activities according to the participant's abilities and progress.
  * Immediate feedback will be provided through the interactive elements of the virtual environment, which increases the child or adolescent's motivation and active participation.
  Interventions: Device: immersive virtual reality intervention with Meta Quest 3
- Control Group (CG): Intervention with Conventional Balance Therapy (Active Comparator): * Participants in the Control Group will receive a standardized conventional physical therapy program focused on balance training.
  * This treatment is based on traditional exercises recognized within pediatric physical therapy to improve postural and functional control in children and adolescents with cerebral palsy.
  * Sessions will also last 30 minutes, three times per week, for six weeks (total: 18 sessions), and will be taught by different pediatric physical therapists than those who treat the Experimental Group, to avoid cross-contamination between groups.
  * Exercises will include:
  Sitting and standing training Balance training on different surfaces Functional activities with manual support or technical aids
  - The goal is to offer an effective therapeutic intervention comparable in time, frequency, and intensity to the Experimental Group, but without the use of VR technology.
  Interventions: Other: Intervention with Conventional Balance Physical Therapy

INTERVENTIONS:
Device: immersive virtual reality intervention with Meta Quest 3 — The intervention consists of a rehabilitation program based on Immersive Virtual Reality (IVR), specifically designed to improve functional balance in children and adolescents with GMFCS levels III and IV cerebral palsy, between 5 and 20 years of age.
  The Meta Quest 3 device will be used, a standalone, wireless, high-definition immersive virtual reality system. This device allows the user to fully immerse themselves in interactive virtual environments, blocking out external stimuli and offering an immersive, motivating, and controlled experience.
  Other Names: virtual reality; meta quest 3; immersive virtual reality
  Arms: Experimental Group (EG): Intervention with Immersive Virtual Reality (VR)
Other: Intervention with Conventional Balance Physical Therapy — The Control Group (CG) will receive a standardized conventional physical therapy program focused on balance training, with the goal of improving postural and functional control in children and adolescents with GMFCS levels III and IV cerebral palsy, between 5 and 20 years of age.
  This treatment is based on traditional exercises recognized within pediatric physical therapy for balance training and is designed to be comparable in time, frequency, and intensity to the experimental group (virtual reality), but without the use of immersive technology.
  Arms: Control Group (CG): Intervention with Conventional Balance Therapy

SUMMARY:
This study proposes a randomized clinical trial to evaluate the effectiveness of an immersive virtual reality (VR)-based rehabilitation intervention on functional balance in children and adolescents (5-20 years) with cerebral palsy (CP), at GMFCS levels III-IV. The experimental group will receive VR therapy using Meta Quest 3 headsets over 6 weeks, compared to a control group receiving conventional balance physiotherapy during the same period. The primary objective is to determine whether VR therapy improves functional balance, assessed using the Early Clinical Assessment of Balance (ECAB). Secondary objectives include evaluating perceived quality of life (PedsQL) and treatment adherence over the 6-week intervention period.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of childhood motor disability, and at GMFCS levels III-IV it involves significant limitations in mobility and balance. Conventional physical therapies have achieved progress in this population but often rely on repetitive exercises that may become monotonous, affecting motivation and adherence among children and adolescents. In this context, immersive virtual reality emerges as an innovative rehabilitation tool, offering engaging and playful environments that increase patient motivation. Preliminary evidence suggests that VR provides a safe and stimulating environment that can enhance balance and motor skills in children with CP, although some studies have not found significant differences compared to traditional therapy.

This controlled randomized clinical trial follows international quality standards (CONSORT/SPIRIT guidelines) to ensure methodological rigor and transparency. A total of 40 participants with CP will be recruited and randomly assigned to either the VR intervention or the control group (20 per group). Therapy will be conducted over 6 weeks for both groups, with balance assessments performed by a physiotherapist blinded to the treatment allocation (i.e., unaware whether the participant belongs to the VR or control group). It is anticipated that the immersive VR intervention will significantly improve functional balance (ECAB score) more than conventional therapy. Additionally, improvements in perceived quality of life and high treatment adherence are expected in the VR group. If results confirm these hypotheses, this study would support the incorporation of immersive VR as an effective and safe complementary therapeutic approach in pediatric CP rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age: Children and adolescents between 5 and 20 years old.
* Diagnosis: Medically confirmed diagnosis of cerebral palsy.
* Functional level: Classified as GMFCS (Gross Motor Function Classification System) level III or IV.
* Cognitive ability: Ability to understand basic instructions and participate in interactive activities.
* Medical stability: No uncontrolled seizures in the past 6 months, No recent orthopedic surgeries in the past 6 months, No botulinum toxin administration in the past 3 months, No serious cardiac or respiratory problems that would prevent light exercise.
* Informed consent: Signature of informed consent by a parent or legal guardian.
* Assent of the minor (if applicable): Verbal or written assent from the participant when age or developmentally appropriate.

Exclusion Criteria:

* Severe sensory impairments that interfere with virtual reality (VR): Profound visual impairment (blindness or severely reduced visual acuity that cannot be corrected), severe deafness without compensation through hearing aids (VR relies heavily on visual and auditory stimuli).
* Simultaneous participation in another intensive motor rehabilitation program during the 6-week study period to avoid confounding effects. Standard conventional therapy will be permitted.
* Extreme fear or intolerance to VR technology: If, after a brief initial session, the participant exhibits panic, severe dizziness, or other clear signs of discomfort, they will be excluded for safety and well-being reasons.
* New or uncontrolled medical instability: Any condition that may jeopardize patient safety during the intervention (e.g., acute infections, extreme pain, recent fractures).

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Functional Balance: ECAB Scale (Early Clinical Assessment of Balance) | Week 0 (baseline) Week 7 (post-intervention) Week 13 (follow-up)
  This is a validated scale that assesses postural control in children and adolescents with cerebral palsy. It includes two components:
  * Head and trunk control
  * Balance in sitting and standing Total score: 0 to 100 points, with higher scores indicating better functional balance.
  Assessment by: A physical therapist blinded to the assigned group (independent evaluator).

SECONDARY OUTCOMES:
Perceived Quality of Life: PedsQL 4.0 Questionnaire (cerebral palsy-specific version, in Spanish) | Week 0 (baseline) Week 7 (post-intervention)
  Assesses the participant's subjective perception of their physical, emotional, social, and academic well-being.
  Format: Self-administered by parents or the adolescent, if possible. Total score: Ranges from 0 (very low quality of life) to 100 (high quality of life)

OTHER OUTCOMES:
Treatment Adherence: Attendance and Compliance Record | Diary
  It is measured as the percentage of sessions completed out of the total scheduled (18 total sessions: 3 sessions/week for 6 weeks).
  Objective: To compare adherence between:
  Experimental Group (virtual reality) Control Group (conventional therapy)